CLINICAL TRIAL: NCT01655940
Title: Comparison of the FORE-SITE and INVOS Cerebral Oximeters During Cardiac Surgery
Brief Title: Cerebral Oximeter Comparison Study
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Aymen N Naguib, Director of Pediatric Cardiothoracic Anesthesia, Nationwide Children's Hospital
Other Study IDs: IRB11-00256
Record Dates: First submitted 2011-05-17; First posted 2012-08-02 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Cardiac Bypass Patients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac bypass patients
  Interventions: Device: Somanetics cerebral oximeter; Device: CASMED cerebral oximeter

INTERVENTIONS:
Device: Somanetics cerebral oximeter — Somanetics cerebral oximeter
Device: CASMED cerebral oximeter — CASMED cerebral oximeter

SUMMARY:
In this prospective study to try to standardize the care for patients, the investigators are planning to compare two cerebral oximeters currently in use at NCH in terms of their accuracy in determining the cerebral oxygen saturation as determined by jugular bulb oxygen saturation. Also, the investigators will compare these devices in terms of their response to changes in hemodynamics that occur during cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cardiac bypass patients having surgery at Nationwide Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation | during surgery - Day 1
  cannulation, decannulation, hemodynamic instability

SECONDARY OUTCOMES:
Mean arterial pressure | during surgery - Day 1
  cannulation, decannulation, hemodynamic instability

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States